CLINICAL TRIAL: NCT05547269
Title: Difference in Patient Reported Outcomes and Patellar Tracking Before and After MPFL Reconstruction With or Without Tibial Tuberosity Transposition
Brief Title: PROMs and Patellar Tracking After MPFL Reconstruction With or Without Tibial Tuberosity Transposition
Status: Terminated | Type: Observational
Why Stopped: Due to insufficient participant enrollment. Recruitment significantly lagged behind projections, and a decline in eligible patients at the study site made it unlikely that the study could be successfully completed within a reasonable timeframe.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 4DCT-PROMs-MPFLr
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Patellar Dislocation; Patellar Dislocation, Recurrent; Patellofemoral Maltracking
Keywords: 4DCT; MPFL reconstruction; Patellofemoral instability
MeSH Terms: conditions — Patellar Dislocation; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patellar dislocations cause pain and functional decline in adolescents, which can be restored by a MPFL reconstruction with or without tibial tuberosity transposition. Yet, many reconstruction methods are being used clinically as consensus on the ideal MPFL reconstruction method is lacking. We propose a soft-tissue loop reconstruction method which potentially decreases the risk for of iatrogenic fracture of the patella and prevents femoral tunnel malposition.

DETAILED DESCRIPTION:
Rationale: A patellar dislocation is one of the most common acute knee disorders in children and adolescents, causing pain and functional decline. In order to restore healthy kinematics and relieve pain, patients can receive a MPFL reconstruction. Still, there is no consensus on the ideal MPFL reconstruction method. Within the Radboudumc, a dynamic soft-tissue loop method is used for MPFL reconstruction. The method minimizes the risk of iatrogenic fracture of the patella and prevents nonanatomic tracking due to femoral tunnel malposition. Yet, the technique has not been evaluated clinically.

Objective: Evaluate pre- and postoperative reported outcomes in patients receiving an soft tissue loop MPFL reconstruction for the treatment of patellar instability. Additionally, it is aimed to investigate the difference in patella tracking before and ~12 months after surgery measured with 4D CT imaging in patients receiving an MPFL reconstruction with or without TTT for the treatment of patellar instability.

Study design: Prospective single centre observational study.

Study population: 20 patients with recurrent patellofemoral instability who have received or will receive an soft-tissue loop MPFL reconstruction with or without TTT within the Radboudumc.

Main study parameters/endpoints: the main study parameter is the pre- and postoperative difference in patient reported outcome measures (PROMs). The secondary aim is to assess changes in patellar tracking (measured before and 12 months (to ~ 24 months) after surgery).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will undergo a 4D CT scan of their knees after their surgery. Whenever possible, the CT scans will be planned during the regular 12 month check-up appointment day so patients do not have to come separately to the Radboudumc for the CT scan. When the operation was > 12 months ago and patients do have to come to the Radboudumc for the CT scan they will be compensated for their travel expenses with a bol.com gift card of 100 euros. The preoperative 4D CT scan and PROMS that will be used in this study are part of standard care. CT scanning exposes patients to radiation. For this study the level of radiation is estimated as an intermediate level of risk. No additional risks are associated with this study. Potential burdens for patients are predominantly time (for which they will be compensated with a gift card of 100 euros in case they have to come to the Radboudumc for the scan) and additional radiation exposure. No direct personal health benefit is expected. However, the knowledge generated with this study is expected to benefit future patients who need to undergo a MPFL reconstruction with or without TTT.

ELIGIBILITY:
Inclusion Criteria:

* Age of 16 years and older.
* Recurrent patellofemoral instability, for which:

  1. the patient will receive a MPFL reconstruction with or without TTT, or
  2. the patient has received a MPFL reconstruction with or without TTT , on the condition that the patient has a usable preoperative 4D CT scan.
* Informed consent of the patient.

Exclusion Criteria:

* Patients below an age of 16 years.
* Patients that are pregnant.
* BMI > 35
* Patients that are unable to actively flex and extend their knee.
* Patellar stabilizing surgery other than the usual MPFL reconstruction with or without TTT. This includes: trochleoplasty, static MPFL reconstruction, isolated TTT

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 16 years and older with recurrent patellofemoral instability who received a MPFL reconstruction with or without TTT.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported outcomes | 6 weeks preoperative to 6 months postoperative
  Pre- and postoperative difference in patient reported outcome measures (PROMs)
Change in patient-reported outcomes. | 6 weeks preoperative to 12 months postoperative
  Pre- and postoperative difference in patient reported outcome measures (PROMs)

SECONDARY OUTCOMES:
Difference in patellar tracking. | preoperative, 12-~24 months postoperative
  Difference between preoperative and 12-24 months postoperative in patellar tracking. This will be measured with 4D CT imaging and quantified by the patellar tilt and shift. The preoperative 4D CT scan is part of standard care.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands